CLINICAL TRIAL: NCT05805748
Title: Development of a Therapeutic Serious Game in the Rehabilitation of Stroke Patient
Brief Title: Serious Game Therapy in Neglect Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopitaux de Saint-Maurice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NSU-SG 5M
Record Dates: First submitted 2023-03-27; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Unilateral Spatial Neglect
Keywords: rehabilitation; new technology; unilateral spatial neglect
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Each patient was assigned to a group who received 2 rehabilitations for 3 weeks, 1) both serious game training and a conventional rehabilitation first and then conventional rehabilitation alone (group 1, G1), or 2) a conventional rehabilitation first and then both serious game training and a conventional rehabilitation (group 2, G2).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Each patient received 2 rehabilitations : a serious game training and a conventional rehabilitation first (during 3 weeks) and then conventional rehabilitation alone (during 3 weeks)
  Interventions: Behavioral: serious game rehabilitation
- Group 2 (Active Comparator): Each patient received 2 rehabilitations for 3 weeks: a conventional rehabilitation first (during 3 weeks) and then both serious game training and a conventional rehabilitation (during 3 weeks)
  Interventions: Behavioral: serious game rehabilitation

INTERVENTIONS:
Behavioral: serious game rehabilitation — The SG rehabilitation was proposed to be played four times per week for three weeks, for a total of 12 sessions, with 15 min per session (= 60 minutes per week). Conventional rehabilitation comprised five sessions of 45 min of neuropsychological rehabilitation using classical exploration training (= 225 minutes per week).

SUMMARY:
The growing field of new technologies offers new perspectives for neurorehabilitation. Serious games are a promising solution in the rehabilitation of cognitive impairments, and they may be useful in the rehabilitation of unilateral spatial neglect. Investigators developed a rehabilitation program for visual exploration training with a serious game and investigated its efficiency. Twelve patients with unilateral spatial neglect after a right hemispheric stroke were recruited. Six patients assigned to a group received both serious game training and conventional rehabilitation, and after only conventional rehabilitation; and six patients assigned to another group received first conventional rehabilitation and then serious game training and conventional rehabilitation. The investigators compared the two groups after rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral spatial neglect syndrome
* Right cerebral lesion

Exclusion Criteria:

* Epilepsia
* General mental deterioration
* Psychiatric disorder
* No prior history of neurological disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Behavioral Inattention Test (BIT) | up to 6 weeks
  Behavioral Inattention Test (Wilson et al., 1987) (BIT) including the first part of conventional subtests: star and letter cancellation, line crossing, figure and shape copying, line bisection and representational drawing (total score /146)

SECONDARY OUTCOMES:
Catherine Bergego Scale (CBS) | up to 6 weeks
  CBS for therapist (Bergego et al., 1995) is based on the direct observation of the therapist in ten standardised dailylife situations. The score ranges from 0 to 30 (higher scores indicating more severe neglect).
Functional Independence Measure (FIM) | up to 6 weeks
  FIM (Minaire, 1991) is a basic indicator of patient disability. FIM is used to track the changes in the functional ability of a patient during an episode of hospital rehabilitation care.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux de Saint Maurice, Saint-Maurice, France